CLINICAL TRIAL: NCT06817850
Title: Evaluation of the Differences Between Simultaneous SpO2s Readings in the NICU: a Multicenter Observational Study
Brief Title: Neonatal Oximeter Bias Study
Acronym: NOB
Status: Not yet recruiting | Type: Observational
Sponsor: Czech Technical University in Prague (Other)
Collaborators: University Hospital, Motol (Other)
Responsible Party: Sponsor
Other Study IDs: NOB (PRICOIII)
Record Dates: First submitted 2025-01-21; First posted 2025-02-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Respiratory Distress; Oxygenation
Keywords: pulse oximetry; automated FiO2 control; SpO2
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infants in the NICU with two oximeters: Infants in the NICU monitored with two oximeters with probes in preductal locations. The use of A-FiO2 is expected.

SUMMARY:
The study aims to determine if there is a systematic difference (bias) between pulse oximeters used in control systems for automated oxygen delivery (A-FiO2) and those used in monitoring systems.

When using A-FiO2 systems there are commonly two oximeter probes on the infant with two difference readouts. Nurses report frustration that the two readings are often markedly different. It is understandable that physiological differences between sensor sites might reflect different regional oxygen saturation levels. It is also possible that there is a relevant systematic bias between difference monitors and sensors.

Therefore, a large systematic multicenter study is needed to determine whether these frequent differences should be ignored as physiological noise or considered clinically relevant.

DETAILED DESCRIPTION:
The accuracy of clinical pulse oximeters is specified as 3% RMS (root mean squared of the bias and variance) compared to arterial SaO2, in the range of 70-100% SpO2. This combines errors from bias and from scatter (imprecision). These validations are carried out under ideal laboratory conditions; that is, on healthy volunteers who undergo experimental desaturations, and not in the routine clinical environment. In a large multicenter clinical observation study, Ross et al in 2013 identified important related concerns. Specifically, they found that many of the clinical measurements were outside the 3% accuracy envelop. Specifically, they reported that bias varied depending on the level of saturation, the oximeter brand, sensor, race and site perfusion. Others have identified relevant differences in oximeters, oximeter sensors [Maiwald], and skin pigmentation.

Our study would be the first study in the neonatal ICU evaluating bias to consider different oximeters, sensors and sensor sites. It is highly topical in that changes in average SpO2 of 3% have been associated with excess neonatal mortality and morbidity.

This study is planned to investigate the source and magnitude of differences in SpO2 readings from oximeter sensors at different sensor sites that are routinely noticed by clinicians. While these differences are most often ignored and attributed to sensor site perfusion, if systematic they could have marked impact on mortality and morbidity.

The aim of the investigation is to provide practical guidance relating to SpO2 bias among oximeters, oximeter sensors and sensor location. While taking advantage of the clinical need for 2 oximeter sensors, the results will be applicable to all neonatal oximeter monitoring.

An observational design was selected to take place in centers using automated FiO2 control systems (A-FiO2) that routinely require the use of one sensor for control and another for monitoring. This is a refinement of the approach used in the often-cited multicenter evaluation of neonatal SpO2 exposure. Thus, without an investigational intervention the observational design is well suited to collect comparable data from multiple centers.

ELIGIBILITY:
Inclusion Criteria:

* Observations of any infant in the neonatal ICU with two simultaneous oximeter monitors may be included. The sites' Ethics Committee must review the protocol, approve participation and determine if Informed Consent is required. If required, it might be prospective, that is prior to collecting any data, or retrospective.

Exclusion Criteria:

* Observations are to be made at the convenience of the Investigative team. They should reflect routine situation, and not be selected to specifically capture problems. Thus, the photo should be taken immediately with both displays are on in the view, and not delayed until something interesting happens. Observations should not be made if any of the following exclusion criteria are meet. If after collection, any of these are meet, the data should not be included as an Observation on the Observation-CRF.

  * One oximeter monitoring post ductal SpO2 in infant with clinically relevant shunt.
  * Monitor and A-FiO2 Oximeter not reading between 70-100%
  * Less than 5 minutes between repeat Observations
  * No more than 5 measurements per day per subject with sensors in same position and same oximeters (i.e., every time either sensor is moved, 5 new Observations can be made that day).
  * Presence of motion artifact
  * Presence of sensor integrity alarms/alerts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants in the NICU monitored with two simultaneous oximeters with probes in preductal locations. The use of A-FiO2 is expected.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Bias between paired SpO2 measurements | 1 month (250 observations is expected from each participating center; on average 2 patients and 5 observations per day per patient assumed)
  Bias between paired SpO2 in three ranges:
  1. Hypoxemia (SpO2: 70 - <89.5%),
  2. Normoxemia (SpO2: 89.5-95.5%)
  3. Hyperoxemia (SpO2: >95.5-100%)
  The ranges are determined as the mean of the two oximeters.

SECONDARY OUTCOMES:
Bias between paired SpO2 related to site | 1 month (250 observations is expected from each participating center; on average 2 patients and 5 observations per day per patient assumed)
  Bias between paired SpO2 (in %) in three ranges related to independent variable: site (as factor).
Bias between paired SpO2 related to sensor location | 1 month (250 observations is expected from each participating center; on average 2 patients and 5 observations per day per patient assumed)
  Bias between paired SpO2 (in %) in three ranges related to independent variable: sensor location (as factor).
Bias between paired SpO2 related to oximeter brand pairs | 1 month (250 observations is expected from each participating center; on average 2 patients and 5 observations per day per patient assumed)
  Bias between paired SpO2 (in %) in three ranges related to independent variable: oximeter brand pairs (as factor).
Bias between paired SpO2 related to sensor pairs | 1 month (250 observations is expected from each participating center; on average 2 patients and 5 observations per day per patient assumed)
  Bias between paired SpO2 (in %) in three ranges related to independent variable: sensor pairs (as factor).
Bias between paired SpO2 related to oximeter averaging setting | 1 month (250 observations is expected from each participating center; on average 2 patients and 5 observations per day per patient assumed)
  Bias between paired SpO2 (in %) in three ranges related to independent variable: oximeter averaging setting (as factor).
Bias between paired SpO2 related to skin shade | 1 month (250 observations is expected from each participating center; on average 2 patients and 5 observations per day per patient assumed)
  Bias between paired SpO2 (in %) in three ranges related to independent variable: skin shade (as factor).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Bachman, MSc, Principal Investigator — Czech Technical University in Prague; Jan Janota, MD, PhD, Principal Investigator — Motol University Hospital
Locations (1):
- Motol University Hospital, Neonatal Unit, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided